CLINICAL TRIAL: NCT01339481
Title: A Phase 0, Open-Label, Multi-Center, Observational Study to Assess the Receptor Occupancy of CD86 and CD80 in Subjects With Rheumatoid Arthritis Initiating Abatacept
Brief Title: A Study to Assess the Receptor Occupancy of CD86 and CD80 in Subjects With Rheumatoid Arthritis Initiating Abatacept
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Perseid Therapeutics LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2408-CL-0103
Record Dates: First submitted 2011-04-13; First posted 2011-04-20 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Orencia; Abatacept; Rheumatoid Arthritis; Infusion
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with RA initiating abatacept treatment regimen: Subjects naïve to both abatacept and belatacept
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept — Intravenous Infusion
  Other Names: Orencia

SUMMARY:
The purpose of this study is to characterize CD86 receptor occupancy in subjects with rheumatoid arthritis (RA) receiving abatacept.

ELIGIBILITY:
Inclusion Criteria:

* Subject has rheumatoid arthritis (RA), is both abatacept- and belatacept-naïve, and is an eligible candidate to start a course of treatment with abatacept in accordance with the product label
* Subject is willing and able to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Rheumatoid Arthritis
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
CD86 Receptor Occupancy | Day 1, Weeks 2, 4, 8, and 12

SECONDARY OUTCOMES:
CD80 Receptor Occupancy | Day 1, Weeks 2, 4, 8, and 12
Abatacept serum concentration | Day 1, Weeks 2, 4, 8 and 12
Change from Day 1 to Week 12 in Subject's Global Assessment of Arthritis | Day 1 and Week 12
Change from Day 1 to Week 12 in Physician's Global Assessment of Arthritis | Day 1 and Week 12
Safety assessed by adverse event reporting including Physical Examination findings | Day 1 through Week 12 post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development; Principal Investigator, Principal Investigator — Metroplex Clinical Research Center
Locations (7):
- United States (7):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arthritis Research of Florida, Palm Harbor, Florida
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - North Shore - Long Island Jewish Health System, Lake Success, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low County Rheumatology, North Charleston, South Carolina
  - Metroplex Clinical Research Center, Dallas, Texas